CLINICAL TRIAL: NCT04285567
Title: A Prospective, Open-Label, Multicenter Randomized Phase III Study to Compare The Efficacy and Safety of A Combined Regimen of Venetoclax and Obinutuzumab Versus Fludarabine, Cyclophosphamide, and Rituximab (FCR)/Bendamustine and Rituximab (BR) in FIT Patients With Previously Untreated Chronic Lymphocytic Leukemia (CLL) Without DEL(17P) or TP53 Mutation
Brief Title: A Study to Compare the Efficacy and Safety of a Combined Regimen of Venetoclax and Obinutuzumab Versus Fludarabine, Cyclophosphamide, and Rituximab (FCR)/ Bendamustine And Rituximab (BR) in FIT Patients With Previously Untreated Chronic Lymphocytic Leukemia (CLL) Without DEL (17P) or TP53 Mutation
Acronym: CRISTALLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO41685; 2019-003327-37 (EudraCT Number); 2023-504036-17-00 (Other: EU CT Number)
Record Dates: First submitted 2020-02-25; First posted 2020-02-26 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; venetoclax; fludarabine; Cyclophosphamide; Rituximab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VEN + G (Experimental): Participants will receive 12 cycles of treatment (each cycle is 28 days). Venetoclax (VEN) will be administered orally, daily, with a 5-week ramp-up period, starting on Cycle 1, Day 22 and administration will continue until the end of Cycle 12. Obinutuzumab (G) will be administered intravenously (IV) on Days 1 (and 2), 8, and 15 of Cycle 1 and on Day 1 of Cycles 2-6.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax
- FCR/BR (Active Comparator): Participants will receive 6 cycles of Fludarabine + Cyclophosphamide + Rituximab (FCR) consisting of a single cycle of a single infusion of rituximab on Day 1 and fludarabine and cyclophosphamide infusions on Days 1-3 of each 28-day cycle or bendamustine (B) as infusions on Days 1 and 2 and a single cycle of rituximab on Day 1 of each 28-day cycle.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab; Drug: Bendamustine

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 milligrams (mg) will be administered IV on Days 1 (and 2), 8, and 15 of Cycle 1 and on Day 1 of Cycles 2-6.
  Other Names: Gazyva; RO5072759; GA101
  Arms: VEN + G
Drug: Venetoclax — Venetoclax 20 mg will be administered orally, once daily starting on Day 22 of Cycle 1 for 7 days, then ramp up from 50 to 400 mg/day during Cycle 2 and continue at 400 mg/day from Day 1 of Cycle 3 till end of Cycle 12.
  Other Names: Venclexta; RO5537382; GDC-0199
  Arms: VEN + G
Drug: Fludarabine — Fludarabine will be administered in a dosage of 25 milligram per meter squared (mg/m^2), IV, on days 1, 2, and 3 of Cycles 1-6.
  Arms: FCR/BR
Drug: Cyclophosphamide — Cyclophosphamide will be administered in a dosage of 250 mg/m^2, IV, on Days 1, 2, and 3 Cycles 1-6.
  Arms: FCR/BR
Drug: Rituximab — Rituximab will be administered at a dose of 375 mg/m^2, IV, on Cycle 1, Day 1 followed by 500 mg/m^2 on Day 1 of Cycles 2-6.
  Other Names: MabThera; Rituxan
  Arms: FCR/BR
Drug: Bendamustine — Bendamustine will be administered at a dose of 90 mg/m^2, IV, on 2 consecutive days of Cycles 1-6.
  Other Names: Treanda; Levact; Ribomustin
  Arms: FCR/BR

SUMMARY:
This study will evaluate the efficacy and safety of venetoclax and obinutuzumab (VEN + G) compared with fludarabine + cyclophosphamide + rituximab or bendamustine + rituximab (FCR/BR) in FIT participants (FIT is defined by a cumulative illness rating scale [CIRS]/score of ≤6 and a normal creatinine clearance of ≥70 mL/min) with previously untreated CLL without DEL(17P) or TP53 mutation requiring treatment. Eligible participants will be randomly assigned in a 1:1 ratio to receive either VEN + G (Arm A) or FCR/BR (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Aged 18 years or older
* Have previously untreated documented Chronic Lymphocytic Leukemia (CLL) according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* CLL requiring treatment according to the iwCLL criteria
* Cumulative Illness Rating Scale (CIRS) score ≤ 6 and creatinine clearance (CrCl) ≥ 70 mL/min
* Hematology values within the following limits, unless cytopenia is caused by the underlying disease (i.e., no evidence of additional bone marrow (BM) dysfunction; e.g., myelodysplastic syndrome, hypoplastic BM):

  * Absolute neutrophil count ≥ 1.0 x 109/L, unless there is BM involvement
  * Platelet count ≥ 75 x 109/L and more than 7 days since last transfusion, or ≥ 30 x 109/L if there is BM involvement
* Adequate liver function as indicated by a total bilirubin, aspartate aminotransferase, and Alanine transaminase ≤ 2 times the institutional upper limit of normal (ULN) value, unless directly attributable to the participant's CLL
* Life expectancy >6 months
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating sperm

Exclusion Criteria:

* Transformation of CLL to aggressive Non-Hodgkin's Lymphoma (NHL)
* Participants with Small Lymphocyclic Lymphoma (SLL) only
* Known central nervous system involvement
* Participants with a history of confirmed progressive multifocal leukoencephalopathy (PML)
* Detected del(17p) or TP53 mutation (valid test within 6-months from screening is required for randomisation)
* An individual organ/system impairment score of 4 as assessed by the Cumulative Illness Rating Scale (CIRS) definition limiting the ability to receive the treatment regimen of this trial with the exception of eyes, ears, nose, throat organ system
* Participants with uncontrolled autoimmune hemolytic anemia or immune thrombocytopenia
* History of prior malignancy
* Participants with infections requiring IV treatment (Grade 3 or 4) within the last 8 weeks prior to enrollment
* Evidence of other clinically significant uncontrolled conditions including but not limited to active or uncontrolled systemic infection (e.g., viral, bacterial, or fungal)
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Hypersensitivity to fludarabine, bendamustine, cyclophosphamide, rituximab, obinutuzumab, or venetoclax or to any of the excipients (e.g., trehalose)
* Pregnant women and nursing mothers
* Vaccination with a live vaccine ≤ 28 days prior to randomization
* Prisoners or participants who are institutionalized by regulatory or court order or persons who are in dependence to the Sponsor or an investigator
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Positive test results for chronic hepatitis B virus (HBV) infection (defined as positive hepatitis B surface antigen [HBsAg] serology)
* Positive test result for hepatitis C (hepatitis C virus [HCV] antibody serology testing)
* Participants with known infection with HIV or Human T-Cell Leukemia Virus 1 (HTLV-1)
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe participation in and completion of the study
* Received any of the following agents within 28 days prior to the first dose of study treatment:

  * Immunotherapy
  * Radiotherapy
  * Hormone therapy
  * Any therapies intended for the treatment of lymphoma/leukemia whether approved or experimental
* Participants who have received the following agents:

  * Strong and moderate CYP3A inhibitors/inducers within 7 days prior to the initiation of study treatment
  * Steroid therapy for anti-neoplastic intent with the exception of inhaled steroids for asthma, topical steroids, or replacement/stress corticosteroids within 7 days prior to the first dose of study drug administration
  * Consumed grapefruit, grapefruit products, Seville oranges(including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of study drug and throughout venetoclax administration
* Inability to swallow a large number of tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2025-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical trial, Study Director — Hoffmann-La Roche
Locations (40):
- United States (4):
  - Medical Center of Aurora, Aurora, Colorado
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - University of Tennessee Medical Center;Office of Clinical Trials, Knoxville, Tennessee
  - Oncology & Hematology Associates of Southwest Virginia, Inc._Goldschmidt, Roanoke, Virginia
- Australia (8):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Liverpool Hospital, Liverpool, New South Wales
  - Port Macquarie - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health;Haematology Research, Clayton, Victoria
  - Peter MacCallum Cancer Centre;Clinical Haematology, Melbourne, Victoria
  - Northern Hospital;Oncology and/or Hematology, Melbourne, Victoria
- France (11):
  - Hopital Haut Leveque Chu de Bordeaux, Pessac, Aquitaine
  - Centre Hospitalier Régional Universitaire de Tours - Hôpital Bretonneau;Hématologie et Thérapie Cellulaire, Tours, Indre-et-Loire
  - Centre Hospitalier de Pérpignan;hématologie, Perpignan, Languedoc-Roussillon
  - Hopital Claude Huriez - CHU de Lille;service maladies appareil digestif, Lille, Nord
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, Provence-Alpes-Côte d'Azur Region
  - centre hospitalier lyon sud;Service Hématologie, Pierre-Bénite, Rhône
  - HENRI MONDOR HOSPITAL;Centre d'investigation clinique, Créteil, Val-de-Marne
  - Centre Hospitalier Universitaire de Caen Normandie, Caen
  - Clinique Victor Hugo- CCS du Mans, Le Mans
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Reims - Hôpital Robert Debré;Hématologie Clinique, Reims
- Italy (10):
  - Instituto Tumori Giovanni Paolo II;ONCOLOGIA MEDICA, Bari, Apulia
  - Ospedale Vito Fazzi;U.O. Ematologia IV Piano Polo Oncologico, Lecce, Apulia
  - Azienda Ospedaliero Universitaria;Ematologia, Modena, Emilia-Romagna
  - Policlinico Umberto I, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Ospedale San Martino;U.O. Clinica Ematologica, Genoa, Liguria
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico;U.O.C Ematologia, Milan, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda;Ematologia, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Maggiore della Carità;SCDU Ematologia, Novara, Piedmont
  - AO Santa Maria della Misericordia, Perugia, Umbria
- Spain (7):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - COMPLEJO HOSPITALARIO DE NAVARRA;Servicio de Hematología, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron;Hematology, Barcelona
  - Hospital Universitario La Paz;Hematología, Madrid
  - Hospital General Universitario Morales Meseguer;Hematologia y Oncologia médica, Murcia
  - Hospital Universitario Virgen del Rocío;Unidad Onco-Hematología Pediátrica, Seville
  - Hospital Universitario de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/innovation/process/clinical-trials/data-sharing).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 166 participants took part in this study which was conducted at 38 investigative sites in France, Italy, Australia, Spain, and the United States. The study is still ongoing.
Pre-assignment Details: Participants with previously untreated chronic lymphocytic leukemia (CLL) without del (17p) or tumor protein p53 (TP53) mutation were randomized in a 1:1 ratio to receive either venetoclax + obinutuzumab (VEN+G) or fludarabine, cyclophosphamide, and rituximab/bendamustine and rituximab (FCR/BR). All participants in FCR/BR arm were eligible for treatment with BR, whereas only participants ≤ 65 years were eligible for FCR. The choice between FCR or BR was at the investigator's discretion.
Groups:
- Arm A: VEN+G: Participants received obinutuzumab, 1000 milligrams (mg), as intravenous (IV) infusion on Days 1 (and 2), 8, and 15 of Cycle 1 and Day 1 of Cycles 2-6. Participants also received venetoclax, with a 5-week ramp-up period (20 mg [Cycle 1 Days 22-28], 50 mg [Cycle 2 Days 1-7], 100 mg [Cycle 2 Days 8-14], 200 mg [Cycle 2 Days 15-21], 400 mg [Cycle 2 Days 22-28]) administered orally, once a day (QD). After the 5-week ramp-up period, participants received venetoclax, 400 mg, orally, QD from Cycle 3 Day 1 until the end of Cycle 12. (1 cycle = 28 days).
- Arm B: FCR/BR: Participants received rituximab (375 milligrams per meter square [mg/m^2] in Cycle 1 and 500 mg/m^2 in Cycles 2-6), on Day 1 of each cycle, plus fludarabine 25 mg/m^2 and cyclophosphamide 250 mg/m^2 on Days 1, 2, and 3 of each cycle as IV infusion up to Cycle 6. Participants alternatively received bendamustine 90 mg/m^2 on Days 1 and 2 of Cycles 1-6 plus rituximab 375 mg/m^2 on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2-6. (1 cycle = 28 days).
Period: Overall Study
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Started | 80 | 86
Safety Population (Safety Population included all participants who received at least one dose of any study medication. Participants were analyzed according to the treatment that they actually received.) | 77 | 85
Completed | 0 | 0
Not Completed | 80 | 86
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Reason Not Specified | 1 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Participants Ongoing in Follow-up | 70 | 74

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants, analyzed according to the treatment to which they were randomized.
Groups:
- Arm A: VEN+G: Participants received obinutuzumab, 1000 mg, as IV infusion on Days 1 (and 2), 8, and 15 of Cycle 1 and Day 1 of Cycles 2-6. Participants also received venetoclax, with a 5-week ramp-up period (20 mg [Cycle 1 Days 22-28], 50 mg [Cycle 2 Days 1-7], 100 mg [Cycle 2 Days 8-14], 200 mg [Cycle 2 Days 15-21], 400 mg [Cycle 2 Days 22-28]) administered orally, QD. After the 5-week ramp-up period, participants received venetoclax, 400 mg, orally, QD from Cycle 3 Day 1 until the end of Cycle 12. (1 cycle = 28 days).
- Arm B: FCR/BR: Participants received rituximab (375 mg/m^2 in Cycle 1 and 500 mg/m^2 in Cycles 2-6), on Day 1 of each cycle, plus fludarabine 25 mg/m^2 and cyclophosphamide 250 mg/m^2 on Days 1, 2, and 3 of each cycle as IV infusion up to Cycle 6. Participants alternatively received bendamustine 90 mg/m^2 on Days 1 and 2 of Cycles 1-6 plus rituximab 375 mg/m^2 on Day 1 of Cycle 1 and 500 mg/m^2 on Day 1 of Cycles 2-6. (1 cycle = 28 days).
- Total: Total of all reporting groups
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR | Total
Number analyzed (Participants) | 80 | 86 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (9.1) | 61.0 (8.6) | 61.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 54
  Male | 55 | 57 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 50 | 62 | 112
  Unknown or Not Reported | 25 | 19 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 58 | 73 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 11 | 31

OUTCOME MEASURES:

1. Primary Outcome: Minimal Residual Disease (MRD) Response Rate Measured in Peripheral Blood (PB) Using Next Generation Sequencing (NGS)
Description: MRD response rate was determined as the percentage of participants with MRD-negativity measured in the PB using NGS using a cutoff of < 10^-4. MRD was considered negative if the result was < 1 CLL cell in 10,000 leukocytes. Percentages have been rounded off to the nearest decimal point.
Time Frame: At Month 15
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 81.3 [70.97 to 89.11] | 54.7 [43.55 to 65.42]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using Cochran-Mantel-Haenszel (CMH) test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Difference in Rates = 26.60, 95% CI 2-sided [12.33 to 40.87] — 95% CI for difference in rates were constructed using Anderson-Hauck method

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first occurrence of disease progression (PD), or death from any cause. PD was assessed by the investigators using the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria. PD was defined as any one of the following: Appearance of any new lesion such as enlarged lymph nodes (≥ 1.5 centimeters [cm]); increase by ≥ 50% in greatest diameter of any previous site (≥ 1.5 cm); increase in the spleen/liver size by ≥ 50% or de novo appearance of splenomegaly/hepatomegaly; increase in blood lymphocytes by 50% or more with at least 5x10^9/litres (L) B lymphocytes; transformation to a more aggressive histology; occurrence of cytopenia; posttreatment: progression of any cytopenia, documented by a decrease of hemoglobin (Hb) ≥ 2 grams per deciliter (g/dL) or 10 g/dL, or by a decrease of platelet counts ≥ 50%/100x10^9/L, which occurs at least 3 months after treatment.
Time Frame: Up to approximately 74 months
Reporting Status: Not Posted, anticipated posting 2027-07

3. Secondary Outcome: MRD Response Rate in PB of FCR/BR Compared With VEN+G at the End of Treatment Response Visit
Description: as for outcome 1
Time Frame: VEN+G: From Cycle 1 Day 1 up to 15 months; FCR/BR: From Cycle 1 Day 1 up to 9 months (1 cycle=28 days)
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 81.3 [70.97 to 89.11] | 60.5 [49.34 to 70.85]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.0053, Cochran-Mantel-Haenszel; Difference in Rates = 20.78, 95% CI 2-sided [6.66 to 34.90] — 95% CI for difference in rates were constructed using Anderson-Hauck method

4. Secondary Outcome: MRD Response Rate in Bone Marrow (BM) of FCR/BR Compared With VEN+G at the End of Treatment Response Visit
Description: MRD response rate=percentage of participants with MRD-negativity measured in BM using NGS (cutoff of <10^-4). MRD negativity=<1 CLL cell in 10,000 leukocytes. MRD in BM was assessed for participants with complete response (CR)/CR with incomplete blood count recovery (CRi) & partial response (PR). CR=PB lymphocytes <4x10^9 /L; Absence of significant lymphadenopathy (nodes <1.5 cm in longest diameter); no hepatomegaly/splenomegaly; absence of disease/constitutional symptoms; BM at least normocellular for age, ≤30% of nucleated cells being lymphocytes. CRi=fulfilling CR criteria but with persistent anemia/thrombocytopenia/neutropenia. PR= ≥50% decrease in PB lymphocyte count from pre-treatment value; ≥50% reduction in lymphadenopathy (sum of longest diameter of up to 6 largest lymph nodes by physical exam & 50% reduction in the sum of product of the diameter of up to 6 largest lymph nodes); ≥50% reduction of liver/spleen enlargement/normalization in size, if enlarged at baseline.
Time Frame: VEN+G: From Cycle 1 Day 1 up to 15 months; FCR/BR: From Cycle 1 Day 1 up to 9 months (1 cycle=28 days)
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized. Percentages have been rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 70.0 [58.72 to 79.74] | 38.4 [28.08 to 49.49]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p < .0001, Cochran-Mantel-Haenszel; Difference in Rates = 31.63, 95% CI 2-sided [16.55 to 46.71] — 95% CI for difference in rates were constructed using Anderson-Hauck method

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with overall response (OR) of CR, CRi, and PR as determined by the investigator according to the iwCLL guidelines. CR was defined as PB lymphocytes <4x10^9 /L; absence of significant lymphadenopathy (nodes <1.5 cm in longest diameter [LD]); no hepatomegaly/splenomegaly; absence of disease/constitutional symptoms; BM at least normocellular for age, ≤30% of nucleated cells being lymphocytes. CRi was defined as fulfilling CR criteria but with persistent anemia/thrombocytopenia/neutropenia. PR was defined as ≥50% decrease in PB lymphocyte count from pre-treatment value; ≥50% reduction in lymphadenopathy sum of longest diameter of up to 6 largest lymph nodes by physical exam and 50% reduction in the sum of product of the diameter of up to 6 largest lymph nodes); ≥50% reduction of liver/spleen enlargement/normalization in size, if enlarged at baseline.
Time Frame: At Month 15
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 88.8 [79.72 to 94.72] | 79.1 [68.95 to 87.10]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.1119, Cochran-Mantel-Haenszel; Difference in Response Rates = 9.68, 95% CI 2-sided [-2.05 to 21.41] — 95% CI for difference in rates were constructed using Anderson-Hauck method

6. Secondary Outcome: CR Rate
Description: CR rate was defined as the percentage of participants with CR or CRi. CR/CRi were defined according to the iwCLL guidelines. CR was defined as one of the following: PB lymphocytes (evaluated by blood and differential count) below 4 x 10^9 /L; absence of significant lymphadenopathy (nodes < 1.5 cm in LD or any extra nodal disease); no hepatomegaly; no splenomegaly; absence of disease or constitutional symptoms; BM at least normocellular for age, ≤30% of nucleated cells being lymphocytes. CRi was defined as participants fulfilling CR criteria but had persistent anemia, thrombocytopenia, or neutropenia. Percentages have been rounded off to the nearest decimal point.
Time Frame: At Month 15
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 50.0 [38.60 to 61.40] | 32.6 [22.84 to 43.52]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.0154, Cochran-Mantel-Haenszel; Difference in Response Rates = 17.44, 95% CI 2-sided [1.96 to 32.93] — 95% CI for difference in rates were constructed using Anderson-Hauck method

7. Secondary Outcome: MRD Response Rate in PB of Participants With a CR/CRi at the End of Treatment Visit
Description: MRD response rate was determined as the percentage of participants (with a CR/CRi) with MRD-negativity measured in the PB using NGS using a cutoff of < 10^-4. MRD was considered negative if the result was < 1 CLL cell in 10,000 leukocytes. CR/CRi were defined according to the iwCLL guidelines. CR was defined as one of the following: PB lymphocytes below 4 x 10^9 /L; absence of significant lymphadenopathy (nodes < 1.5 cm in LD or any extra nodal disease); no hepatomegaly; no splenomegaly; absence of disease or constitutional symptoms; BM at least normocellular for age, ≤30% of nucleated cells being lymphocytes. CRi was defined as participants fulfilling CR criteria but had persistent anemia, thrombocytopenia, or neutropenia. Percentages have been rounded off to the nearest decimal point.
Time Frame: At Month 15
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized. Overall number analyzed is the number of participants with CR/CRi.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 40 | 28
percentage of participants | 97.5 [86.84 to 99.94] | 78.6 [59.05 to 91.70]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.0054, Cochran-Mantel-Haenszel; Difference in Rates = 18.93, 95% CI 2-sided [0.91 to 36.95] — 95% CI for difference in rates were constructed using Anderson-Hauck method

8. Secondary Outcome: MRD Response Rate in BM of Participants With a CR/CRi at the End of Treatment Visit
Description: MRD response rate was determined as the percentage of participants (with CR/CRi) with MRD-negativity measured in the BM using NGS using a cutoff of < 10^-4. MRD was considered negative if the result was < 1 CLL cell in 10,000 leukocytes. CR/CRi were defined according to the iwCLL guidelines. CR was defined as one of the following: PB lymphocytes below 4 x 10^9 /L; absence of significant lymphadenopathy (nodes < 1.5 cm in LD or any extra nodal disease); no hepatomegaly; no splenomegaly; absence of disease or constitutional symptoms; BM at least normocellular for age, ≤30% of nucleated cells being lymphocytes. CRi was defined as participants fulfilling CR criteria with CR but had persistent anemia, thrombocytopenia, or neutropenia. Percentages have been rounded off to the nearest decimal point.
Time Frame: VEN+G: From Cycle 1 Day 1 up to 15 months; FCR/BR: From Cycle 1 Day 1 up to 9 months (1 cycle=28 days)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 40 | 28
percentage of participants | 87.5 [73.20 to 95.81] | 60.7 [40.58 to 78.50]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.0038, Cochran-Mantel-Haenszel; Difference in Rates = 26.79, 95% CI 2-sided [3.86 to 49.72] — 95% CI for difference in rates were constructed using Anderson-Hauck method

9. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented OR (CR, CRi and PR) to the time of PD as determined by the investigator, or death from any cause, whichever occurs first. CR, CRi, PR, and PD were defined according to the iwCLL guidelines. PD was defined as any one of the following: appearance of any new lesion such as enlarged lymph nodes (≥ 1.5 cm); increase by ≥ 50% in greatest diameter of any previous site (≥ 1.5 cm); increase in the spleen/liver size by ≥ 50% or de novo appearance of splenomegaly/hepatomegaly; increase in blood lymphocytes by 50% or more with at least 5x10^9/L B lymphocytes; transformation to a more aggressive histology; occurrence of cytopenia; posttreatment: progression of any cytopenia, documented by a decrease of Hb ≥ 2 g/dL or 10 g/dL, or by a decrease of platelet counts ≥ 50%/100x10^9/L, which occurs at least 3 months after treatment. CR, CRi and PR were defined as outlined in the description for ORR outcome measure (OM) number 5.
Time Frame: Up to approximately 74 months
Reporting Status: Not Posted, anticipated posting 2027-07

10. Secondary Outcome: Best Overall Response (BOR)
Description: BOR=percentage of participants with CR/CRi/PR/stable disease (SD)/PD per the investigator. Participants with best response as CR/CRi/PR were considered responders while those reaching SD/PD were non-responders. SD=participants who have not achieved a CR or a PR, or who have not exhibited PD. PD=any one of the following: appearance of any new lesion such as enlarged lymph nodes (≥ 1.5 cm); increase by ≥ 50% in greatest diameter of any previous site (≥ 1.5 cm); increase in the spleen/liver size by ≥ 50% or de novo appearance of splenomegaly/hepatomegaly; increase in blood lymphocytes by 50% or more with at least 5x10^9/L B lymphocytes; transformation to a more aggressive histology; occurrence of cytopenia; posttreatment: progression of any cytopenia, documented by a decrease of Hb ≥ 2 g/dL or 10 g/dL, or by a decrease of platelet counts ≥ 50%/100x10^9/L, which occurs at least 3 months after treatment. CR, CRi and PR were defined as outlined in the description for ORR, OM number 5.
Time Frame: At Month 15
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
Number analyzed (Participants) | 80 | 86
percentage of participants | 93.8 [86.01 to 97.94] | 90.7 [82.49 to 95.90]
Statistical Analysis 1: Comparison: Arm A: VEN+G vs Arm B: FCR/BR; P-value estimated using CMH test stratified by the IvRS randomization stratification factors; Test type: Superiority; p = 0.4199, Cochran-Mantel-Haenszel; Difference in Response Rates = 3.05, 95% CI 2-sided [-5.73 to 11.84] — 95% CI for difference in rates were constructed using Anderson-Hauck method

11. Secondary Outcome: Event-free Survival (EFS)
Description: EFS was defined as the time between the date of randomization and the date of PD/relapse, death, or the start of a new anti-leukemic therapy. PD was defined as any one of the following: appearance of any new lesion such as enlarged lymph nodes (≥ 1.5 cm); increase by ≥ 50% in greatest diameter of any previous site (≥ 1.5 cm); increase in the spleen/liver size by ≥ 50% or de novo appearance of splenomegaly/hepatomegaly; increase in blood lymphocytes by 50% or more with at least 5x10^9/L B lymphocytes; transformation to a more aggressive histology; occurrence of cytopenia; posttreatment: progression of any cytopenia, documented by a decrease of Hb ≥ 2 g/dL or 10 g/dL, or by a decrease of platelet counts ≥ 50%/100x10^9/L, which occurs at least 3 months after treatment.
Time Frame: Up to approximately 74 months
Reporting Status: Not Posted, anticipated posting 2027-07

12. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time between the date of randomization and the date of death due to any cause.
Time Frame: Up to approximately 74 months
Reporting Status: Not Posted, anticipated posting 2027-07

13. Secondary Outcome: VEN + G: Tumor Lysis Syndrome (TLS) Risk Reduction Rate
Description: TLS risk reduction rate in the VEN + G arm was defined as the reduction in the percentage of participants who were TLS high-risk after 3 doses of obinutuzumab compared to the percentage of participants who were TLS high-risk at baseline. Risk for developing TLS were categorised into: Low - All measurable lymph nodes with the LD < 5 cm and < 25x10^9/L absolute lymphocyte count (ALC); Medium - Any measurable lymph node with the LD ≥5 cm but <10 cm OR ≥25x10^9/L ALC; High - Any measurable lymph node with the LD ≥10 cm or the presence of both ≥25x10^9/L ALC and any measurable lymph node with the LD ≥5 cm but <10 cm. Percentages have been rounded off to the nearest decimal point.
Time Frame: Baseline up to Cycle 1 Day 22 (1 cycle=28 days)
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: VEN+G
Number analyzed (Participants) | 80
percentage of participants
  High-risk at Baseline | 23.8
  High-risk at Cycle 1 Day 22 | 0

14. Secondary Outcome: VEN + G: Reduction in Mandatory Hospitalizations During Venetoclax Ramp-up
Description: Reduction in mandatory hospitalizations during venetoclax ramp-up in the VEN + G arm participants was defined as the actual number of protocol-mandated hospitalizations for TLS monitoring during venetoclax ramp-up period after 3 doses of obinutuzumab compared to the number of protocol-mandated hospitalizations for TLS monitoring during venetoclax ramp-up expected at baseline. Ramp-up period for venetoclax was defined as period from Cycle 1, Days 22-28, and Cycle 2, Day 1-Day 7 where the 20 mg and 50 mg daily doses of venetoclax, were administered for participants at TLS-high risk requiring mandated hospitalizations (the hospitalizations at 100, 200 and 400 was only needed if the participant had a TLS event at one of the lower doses). Total number of hospitalizations in high-risk TLS participants at baseline (expected to be N=2 hospitalization) was compared with the number of protocol mandated hospitalizations during the first 2 doses of the ramp-up.
Time Frame: Cycle 1 Days 22-28 up to Cycle 2 Days 1-7 (1 cycle=28 days)
Population: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
Measure: Number; unit: number of hospitalizations
Arm/Group | Arm A: VEN+G
Number analyzed (Participants) | 80
number of hospitalizations | 2

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was any AE that meets any of the following criteria: is fatal; is life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug; is a significant medical event in the investigator's judgment.
Time Frame: From Day 1 until 28 days after the last dose of study drug, or until initiation of another anti-cancer therapy (up to 74 months)
Reporting Status: Not Posted, anticipated posting 2027-07

16. Secondary Outcome: Number of Participants With Premature Withdrawals Due to AEs
Description: as for outcome 15
Time Frame: as for outcome 15
Reporting Status: Not Posted, anticipated posting 2027-07

17. Secondary Outcome: Change From Baseline in Physical Functioning, Role Functioning and Health-Related Quality of Life (HRQoL) Assessed Using European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30 (EORTC QLQC-30)
Description: The EORTC QLQ-C30 consists of 30 questions incorporated into five functional scales (physical, role, cognitive, emotional and social scales), three symptom scales (fatigue, pain, nausea, and vomiting scales), a global health status/global quality-of-life (GHS/QoL) scale, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The 28 function and symptom items were scored on a 4-point scale that ranged from "not at all" to "very much," and the 2 GHS/QoL items were scored on a 7-point scale that ranged from "very poor" to "excellent." Raw average scale scores were linearly transformed to range 0-100 with higher scores indicating higher response levels (i.e. higher functioning, higher symptom severity).
Time Frame: VEN + G: Day 1 of Cycle 1-12, Day 28 after treatment completion/early termination (TC/ET), follow up (FU) visits; FCR/BR: Day 1 of Cycle 1-6, Day 28 after TC/ET, end of combination treatment response visit and FU visit (up to 74 months) (1 cycle=28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

18. Secondary Outcome: Change From Baseline in M.D. Anderson Symptom Inventory-CLL (MDASI-CLL) Score
Description: MDASI-CLL consists of 25 items over 3 scales that assess core cancer & CLL-related symptom severity, as well as symptom interference that a participant may have experienced in past 24 hours. Participants were asked to rate severity of 13 symptoms called mean core symptom severity (pain, fatigue, nausea, disturbed sleep, distressed, shortness of breath, remembering things, lack of appetite, drowsy, dry mouth, sadness, vomiting & numbness/tingling), 6 disease-specific symptoms called mean module symptom severity (night sweats, fever & chills, lymph node swelling, diarrhea, easy bruising/bleeding & constipation) & 6 mean interference on life questions (general activity, walking, work, mood, relations with other people & enjoyment of life) on a scale from 0-10 with 0 indicating that symptom is "not present" or "did not interfere" with participant's activities & 10 indicating "as bad as you can imagine" or "interfered completely". Lower scores indicated lower symptom severity/interference.
Time Frame: VEN + G: Day 1 of Cycle 1-12, Day 28 after TC/ET, FU visits; FCR/BR: Day 1 of Cycle 1-6, Day 28 after TC/ET, end of combination treatment response visit and FU visit (up to approximately 74 months) (1 cycle=28 days)
Reporting Status: Not Posted, anticipated posting 2027-07

ADVERSE EVENTS:
Time Frame: Up to approximately 44.4 months
Description: AEs: Safety Population included all participants who received at least one dose of any study medication.
  All-cause mortality: FAS included all randomized participants, analyzed according to the treatment to which they were randomized.
  This study is ongoing and data collected up to the primary completion date are reported here. AE data will be updated one year after study completion date.
Arm/Group | Arm A: VEN+G | Arm B: FCR/BR
All-Cause Mortality (participants affected / at risk) | 3/80 | 3/86
Serious Adverse Events (participants affected / at risk) | 47/77 | 42/85
Other Adverse Events (participants affected / at risk) | 76/77 | 80/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: VEN+G (N=77) | Arm B: FCR/BR (N=85)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 7 (11)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Apical granuloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 9 (11)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Beta haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (9) | 6 (7)
COVID-19 pneumonia (Infections and infestations) | 7 (8) | 5 (5)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Pneumonia fungal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 4 (4)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (10) | 6 (6)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 3 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypouricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Eccrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease lymphocyte predominance type stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: VEN+G (N=77) | Arm B: FCR/BR (N=85)
Anaemia (Blood and lymphatic system disorders) | 13 (21) | 12 (14)
Neutropenia (Blood and lymphatic system disorders) | 43 (106) | 40 (81)
Thrombocytopenia (Blood and lymphatic system disorders) | 30 (41) | 18 (24)
Tachycardia (Cardiac disorders) | 4 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 19 (20)
Diarrhoea (Gastrointestinal disorders) | 27 (32) | 11 (14)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 16 (19) | 34 (67)
Vomiting (Gastrointestinal disorders) | 4 (6) | 19 (25)
Asthenia (General disorders) | 10 (12) | 11 (13)
Chills (General disorders) | 3 (3) | 5 (5)
Fatigue (General disorders) | 9 (13) | 15 (17)
Pyrexia (General disorders) | 14 (17) | 10 (13)
COVID-19 (Infections and infestations) | 32 (35) | 25 (29)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2)
Incorrect drug administration rate (Injury, poisoning and procedural complications) | 0 (0) | 5 (13)
Infusion related reaction (Injury, poisoning and procedural complications) | 50 (80) | 34 (51)
Alanine aminotransferase increased (Investigations) | 5 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 4 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (12) | 6 (10)
Platelet count decreased (Investigations) | 4 (5) | 5 (8)
White blood cell count decreased (Investigations) | 0 (0) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (8) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (12) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 2 (3)
Headache (Nervous system disorders) | 8 (9) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 2 (2)
Insomnia (Psychiatric disorders) | 7 (7) | 6 (6)
Dysuria (Renal and urinary disorders) | 1 (1) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 23 (27)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 7 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/67/NCT04285567/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT04285567/SAP_001.pdf